CLINICAL TRIAL: NCT06696014
Title: MIrikizumab in UC - a Real-woRld prOspective multicenteR Registry
Brief Title: Mirikizumab Real World Protocol
Acronym: MIRROR
Status: Recruiting | Type: Observational
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Other Study IDs: 24-2191
Record Dates: First submitted 2024-11-11; First posted 2024-11-19 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-07

CONDITIONS: Ulcerative Colitis
Keywords: mirikizumab; Omvoh; MIRROR
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 52 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to learn about how effective mirikizumab (Omvoh) is when treating patients with ulcerative colitis (UC)

Does mirikizumab (Omvoh) lead to a reduction in symptoms at intervals throughout one year?

Participants being prescribed mirikizumab (Omvoh) as part of their regular medical care for UC will answer online survey questions about their bowel habits for 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, age 18 years or older, with UC, who within 2 weeks have been started on mirikizumab therapy for moderate to severe UC or who plan to begin this therapy within the next 2 weeks. The start of the mirikizumab treatment must have been or be initiated in the setting of standard-of-care therapy.
* Anticipation that the patient will be followed by the participating center for the next 12 months.
* Diagnosis of UC must be established based on standard clinical, radiographic, endoscopic, and histologic criteria as described below.

Criteria for diagnosis of UC The following diagnostic criteria were developed by the NIDDK IBD Genetics Consortium and are provided as guidelines to complete documentation on individuals with Ulcerative Colitis.

A) Symptoms including one or more: diarrhea, rectal bleeding, abdominal pain, fever, extraintestinal manifestations, weight loss, or failure to thrive.

AND

B) Symptoms on two or more occasions separated by at least 8 weeks or ongoing symptoms of at least 6 weeks duration.

AND

C) Endoscopic Findings compatible with UC:

* Superficial inflammation and/or ulceration (involving only the mucosa and submucosa) of the colon, which is continuous from the rectum extending proximally without skip lesions or complete rectal sparing (relative rectal sparing is allowed for patients receiving topical, rectal therapy; patchiness of endoscopic inflammation may be observed in patients with partially treated ulcerative colitis).
* In patients with proctitis or left-sided ulcerative colitis, there may be an area of inflammation in the cecum, usually surrounding the appendiceal orifice.
* No inflammation of the small intestine ("backwash ileitis" is allowed - non-stenotic superficial inflammation of the terminal ileal mucosa associated with severe pancolitis, which resolves following medical or surgical treatment of the colitis).
* No features of Crohn's disease listed above. There is no minimum length of extension of UC required for inclusion in this study.

Exclusion Criteria:

Patients will be excluded if they meet any of the following criteria:

* Inability to provide informed consent.
* Non-English speaking.
* Patients presenting for a one-time consultation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with ulcerative colitis starting mirikizumab in the setting of standard-of-care
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-05-08 (Actual); Primary Completion 2030-01-01 (Estimated); Study Completion 2030-01 (Estimated)

PRIMARY OUTCOMES:
induction of clinical response as evaluated by the Simple Clinical Colitis Activity Index (SCCAI) for the patient-reported outcomes. | Weeks 1,2,4,8,12,18,24,36, and 52 after the start of therapy (each time point will be assessed separately)
  The SCCAI is a 6-item that describes the symptoms and disease activity of a patient with UC at the time of assessment. A score of 0-4 is considered a clinical range of remission (but with more refined definitions of clinical remission with SCCAI ≤2 and very mild symptoms with a score >2 ≤4), 5-7 mild activity, 8-16 moderate activity and > 16 severe activity.
  A response will be defined as a decrease of the SCCAI score < 5 points in patients with a baseline SCCAI ≥5.

SECONDARY OUTCOMES:
Remission as measured by Patient-Reported Outcomes Measurement Information System (PROMIS)-Depression Scoreoint will be assessed separately) (as measured by various PROs as outlined in methods) | Weeks 0, 12, 24, and 52.
  Description: PROMIS measure of depression measures well-being. This is calculated as T scores. A clinically meaningful difference is considered to be a change in T score of ≥ 2.5 (scores are normalized at 50 with a standard deviation of 10). Differences in PROMIS scores compared to baseline will be assessed.
Remission as measured by PROMIS-Anxiety Score | Weeks 0, 12, 24, and 52
  PROMIS measure of anxiety measures well-being. This is calculated as T scores. A clinically meaningful difference is considered to be a change in T score of ≥ 2.5 (scores are normalized at 50 with a standard deviation of 10). Differences in PROMIS scores compared to baseline will be assessed.
Remission as measured by PROMIS-Sleep Score | Weeks 0, 12, 24, and 52
  PROMIS measure of sleep measures well-being. This is calculated as T scores. A clinically meaningful difference is considered to be a change in T score of ≥ 2.5 (scores are normalized at 50 with a standard deviation of 10). Differences in PROMIS scores compared to baseline will be assessed.
Remission as measured by PROMIS-Social Satisfaction Score | Weeks 0, 12, 24, and 52
  PROMIS measure of satisfaction measures well-being. This is calculated as T scores. A clinically meaningful difference is considered to be a change in T score of ≥ 2.5 (scores are normalized at 50 with a standard deviation of 10). Differences in PROMIS scores compared to baseline will be assessed.
Remission as measured by Likert scale urgency Score | Weeks 1,2,4,8,12,18,24,36, and 52 after the start of therapy
  Urgency will be measured by the 11-point Likert scale urgency question as validated in the mirikizumab clinical trials. Score range is 0-10. The higher the score, the worse the urgency.
Remission as measured by Functional Assessment of Chronic Illness Therapy (FACIT)- Fatigue Scale Score | Baseline (Week 0), Weeks 12, 24, and 52
  Fatigue will be determined by the validated FACIT-F questionnaire. The FACIT-F is a 13-item measure that assesses self-reported fatigue and its impact upon daily activities and function. Score range is 0-52. The higher the score, the better the quality of life.
Remission as measured by The Short Inflammatory Bowel Disease Questionnaire (SIBDQ) score | Weeks 0,4,8,12,18,24,36 and 52
  The SIBDQ is a disease-specific health-related quality of life (HRQOL) questionnaire, able to detect and define meaningful clinical changes in inflammatory bowel disease (IBD) participants by measuring physical, social and emotional status. The SIBDQ consists of 10 questions; each question is scored on a scale from 1 (poor QOL) to 7 (optimum QOL). A higher score indicates a better health-related quality of life. Total scores range from 10 (poor QoL) to 70 (good QoL).

CONTACTS AND LOCATIONS:
Overall Officials: Hans Herfarth, MD, PhD, Principal Investigator — University of North Carolina
Locations (9):
- United States (8):
  - South Denver Gastroenterology, Denver, Colorado
  - AdventHealth, Orlando, Florida
  - University of Iowa Health Care, Iowa City, Iowa
  - University of Louisville, Clinical Trials Unit, Louisville, Kentucky
  - University Of Rochester Medical Center, Rochester, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - Medical University of South Carolina (MUSC), Charleston, South Carolina
  - Southern Star Research Institute, LLC, San Antonio, Texas
- TIDHI Innovation Inc., Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared beginning 3 to 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with the University of North Carolina [UNC].
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Beginning 3 months and ending 36 months following article publication.
Access Criteria: Researchers who provide a methodologically sound proposal.

REFERENCES:
- [Result] Dubinsky M, Bleakman AP, Panaccione R, Hibi T, Schreiber S, Rubin D, Dignass A, Redondo I, Gibble TH, Kayhan C, Travis S. Bowel Urgency in Ulcerative Colitis: Current Perspectives and Future Directions. Am J Gastroenterol. 2023 Nov 1;118(11):1940-1953. doi: 10.14309/ajg.0000000000002404. Epub 2023 Jun 12. PMID 37436151
- [Result] Singh S, Ananthakrishnan AN, Nguyen NH, Cohen BL, Velayos FS, Weiss JM, Sultan S, Siddique SM, Adler J, Chachu KA; AGA Clinical Guidelines Committee. Electronic address: clinicalpractice@gastro.org. AGA Clinical Practice Guideline on the Role of Biomarkers for the Management of Ulcerative Colitis. Gastroenterology. 2023 Mar;164(3):344-372. doi: 10.1053/j.gastro.2022.12.007. PMID 36822736
- [Result] Higgins PD, Schwartz M, Mapili J, Krokos I, Leung J, Zimmermann EM. Patient defined dichotomous end points for remission and clinical improvement in ulcerative colitis. Gut. 2005 Jun;54(6):782-8. doi: 10.1136/gut.2004.056358. PMID 15888785
- [Result] Barnes EL, Hanson JS, Regueiro MD, Saha S, Sands BE, Rubin DT, Dubinsky MC, Siegel CA, Gazis DR, Crawford JM, Long MD. Older Adult Patients Use More Aminosalicylate Monotherapy Compared With Younger Patients With Inflammatory Bowel Disease: TARGET-IBD. J Clin Gastroenterol. 2022 Jul 1;56(6):529-535. doi: 10.1097/MCG.0000000000001557. Epub 2021 Jun 11. PMID 34115661
- [Result] Tinsley A, Macklin EA, Korzenik JR, Sands BE. Validation of the functional assessment of chronic illness therapy-fatigue (FACIT-F) in patients with inflammatory bowel disease. Aliment Pharmacol Ther. 2011 Dec;34(11-12):1328-36. doi: 10.1111/j.1365-2036.2011.04871.x. Epub 2011 Oct 17. PMID 21999576
- [Result] Dubinsky MC, Clemow DB, Hunter Gibble T, Li X, Vermeire S, Hisamatsu T, Travis SPL. Clinical Effect of Mirikizumab Treatment on Bowel Urgency in Patients with Moderately to Severely Active Ulcerative Colitis and the Clinical Relevance of Bowel Urgency Improvement for Disease Remission. Crohns Colitis 360. 2022 Dec 13;5(1):otac044. doi: 10.1093/crocol/otac044. eCollection 2023 Jan. PMID 36777368
- [Result] Outtier A, Gijbels L, Noman M, Verstockt B, Sabino J, Vermeire S, Ferrante M. Screening Failure in a Large Clinical Trial Centre for Inflammatory Bowel Diseases: Rates, Causes, and Outcomes. Inflamm Bowel Dis. 2023 Sep 1;29(9):1440-1445. doi: 10.1093/ibd/izac227. PMID 36350998
- [Result] Bewtra M, Brensinger CM, Tomov VT, Hoang TB, Sokach CE, Siegel CA, Lewis JD. An optimized patient-reported ulcerative colitis disease activity measure derived from the Mayo score and the simple clinical colitis activity index. Inflamm Bowel Dis. 2014 Jun;20(6):1070-8. doi: 10.1097/MIB.0000000000000053. PMID 24810138
- [Result] Long MD, Afzali A, Fischer M, Hudesman D, Abdalla M, McCabe R, Cohen BL, Ungaro RC, Harlan W, Hanson J, Konijeti G, Polyak S, Ritter T, Salzberg B, Seminerio J, English E, Zhang X, Sharma PP, Herfarth HH. Tofacitinib Response in Ulcerative Colitis (TOUR): Early Response After Initiation of Tofacitinib Therapy in a Real-world Setting. Inflamm Bowel Dis. 2023 Apr 3;29(4):570-578. doi: 10.1093/ibd/izac121. PMID 35700276
- [Result] Ha C, Ullman TA, Siegel CA, Kornbluth A. Patients enrolled in randomized controlled trials do not represent the inflammatory bowel disease patient population. Clin Gastroenterol Hepatol. 2012 Sep;10(9):1002-7; quiz e78. doi: 10.1016/j.cgh.2012.02.004. Epub 2012 Feb 15. PMID 22343692
- [Result] Dulai PS, Singh S, Jairath V, Wong E, Narula N. Integrating Evidence to Guide Use of Biologics and Small Molecules for Inflammatory Bowel Diseases. Gastroenterology. 2024 Mar;166(3):396-408.e2. doi: 10.1053/j.gastro.2023.10.033. Epub 2023 Nov 8. PMID 37949249
- [Result] Lichtenstein GR, Yan S, Bala M, Hanauer S. Remission in patients with Crohn's disease is associated with improvement in employment and quality of life and a decrease in hospitalizations and surgeries. Am J Gastroenterol. 2004 Jan;99(1):91-6. doi: 10.1046/j.1572-0241.2003.04010.x. PMID 14687148
- [Result] Ananthakrishnan AN, Weber LR, Knox JF, Skaros S, Emmons J, Lundeen S, Issa M, Otterson MF, Binion DG. Permanent work disability in Crohn's disease. Am J Gastroenterol. 2008 Jan;103(1):154-61. doi: 10.1111/j.1572-0241.2007.01561.x. Epub 2007 Dec 11. PMID 18076736
- [Result] Shivashankar R, Tremaine WJ, Harmsen WS, Loftus EV Jr. Incidence and Prevalence of Crohn's Disease and Ulcerative Colitis in Olmsted County, Minnesota From 1970 Through 2010. Clin Gastroenterol Hepatol. 2017 Jun;15(6):857-863. doi: 10.1016/j.cgh.2016.10.039. Epub 2016 Nov 14. PMID 27856364
- [Result] Herrinton LJ, Liu L, Lewis JD, Griffin PM, Allison J. Incidence and prevalence of inflammatory bowel disease in a Northern California managed care organization, 1996-2002. Am J Gastroenterol. 2008 Aug;103(8):1998-2006. doi: 10.1111/j.1572-0241.2008.01960.x. PMID 18796097
- [Result] Loftus EV Jr, Schoenfeld P, Sandborn WJ. The epidemiology and natural history of Crohn's disease in population-based patient cohorts from North America: a systematic review. Aliment Pharmacol Ther. 2002 Jan;16(1):51-60. doi: 10.1046/j.1365-2036.2002.01140.x. PMID 11856078